CLINICAL TRIAL: NCT01814371
Title: Individualized vs. Household Eradication of MRSA in Households With Children
Brief Title: Individualized vs. Household MRSA Decolonization
Acronym: HOME2DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Stephanie A. Fritz, Assistant Professor of Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HS021736 (AHRQ)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Staphylococcal Skin Infection; Abscess; Furunculosis; Staphylococcus Aureus; MRSA Infection
Keywords: Abscesses; Furunculosis; Staphylococcus aureus colonization; Staphylococcal Skin Infection; MRSA
MeSH Terms: conditions — Staphylococcal Skin Infections; Abscess; Furunculosis; Staphylococcal Infections | interventions — Mupirocin; Indicator Dilution Techniques; Sodium Hypochlorite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized Approach (Active Comparator): The decolonization regimen will be performed only by those household members who experienced SSTI in the prior year.
  Interventions: Drug: 2% mupirocin ointment; Other: Bleach Bath (dilute); Behavioral: Hygiene Protocol
- Household Approach (Active Comparator): All members of the household will perform the decolonization regimen.
  Interventions: Drug: 2% mupirocin ointment; Other: Bleach Bath (dilute); Behavioral: Hygiene Protocol

INTERVENTIONS:
Drug: 2% mupirocin ointment — Participants over 1 month of age, apply ointment to the anterior nares twice daily for 5 days.
  Other Names: Bactroban
Other: Bleach Bath (dilute) — Participants over 1 month of age, pour 1/4 cup of bleach into a bath tub filled 1/4 full of water. Soak in bath for 15 minutes daily for 5 days.
  Other Names: Clorox
Behavioral: Hygiene Protocol — Follow key hygiene tips:
  * Throw out all lotions or creams that you dip your hands into and replace with pumps or pour bottles.
  * Use liquid(pour or pump) soaps instead of bar soaps.
  * Wash hands frequently or use hand sanitizer(with more than %60 alcohol) such as Germ-X or Purell.
  * Do not share personal care items such as razors, brushes, or deodorant.
  * Wash all sheets and towels in hot water. Wash sheets every week.
  * Use towels and wash cloths only once before washing and do not share.

SUMMARY:
The purpose of this research study is to compare the effectiveness of commonly used decolonization treatments (application of mupirocin antibiotic ointment to the nose and bleach baths) when performed by individuals with a history of skin and soft tissue infection (SSTI) in the prior year (individualized approach) in comparison to decolonization of all household members (household approach) in an attempt to prevent Staphylococcus aureus skin infections. The investigators hypothesize an individualized decolonization approach will be equally as effective as a household approach to prevent SSTI.

DETAILED DESCRIPTION:
Methicillin-resistant Staphylococcus aureus (MRSA) was once uniformly associated with hospital-acquired infections; however, MRSA strains have emerged that thrive outside the hospital environment, causing significant morbidity and mortality among immunocompetent individuals, leading to their designation as community-acquired methicillin resistant Staphylococcus aureus (CA-MRSA).

There is no available vaccine against S. aureus. Thus, other preventive measures, including topical antimicrobial therapies, have been used in an attempt to prevent staphylococcal infections. These therapies include mupirocin (a topical antibiotic with activity against MRSA) and dilute bleach water baths. The effectiveness of these measures directed at patients colonized with traditional MSSA and HA-MRSA strains in an attempt to prevent nosocomial infections varies across studies, and maintenance of eradication diminishes over time. With the emergence of the CA-MRSA epidemic, these measures have been extrapolated to patients in community settings. We aim to find a practical approach to decolonization which patients can feasibly perform at home to reduce the incidence of skin and soft tissue infections(SSTI).

Specific Aim: Compare the effectiveness of decolonization of individuals with a history of SSTI in the prior year (individualized approach) to decolonization of all household members (household approach) in reducing the incidence of recurrent SSTI. Primary hypothesis: An individualized decolonization approach will be equally as effective as decolonization of all household members to prevent SSTI. Secondary hypothesis: Application of mupirocin to the anterior nares twice daily for 5 days will not result in a higher prevalence of colonization with mupirocin-resistant strains at subsequent longitudinal samplings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are enrolled in a 12-month observational study entitled "The Community-Associated Methicillin-Resistant Staphylococcus aureus Among Household Members and the Home Environment Study."

Exclusion Criteria:

* Households in which all members experienced SSTI during the 12-month observational study
* Individuals with known allergies to mupirocin or bleach (sodium hypochlorite)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2013-04; Primary Completion 2017-02-26 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Fritz, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Hogan PG, Parrish KL, Mork RL, Boyle MG, Muenks CE, Thompson RM, Morelli JJ, Sullivan ML, Hunstad DA, Bubeck Wardenburg J, Rzhetsky A, Gehlert SJ, Burnham CD, Fritz SA. HOME2 Study: Household Versus Personalized Decolonization in Households of Children With Methicillin-Resistant Staphylococcus aureus Skin and Soft Tissue Infection-A Randomized Clinical Trial. Clin Infect Dis. 2021 Dec 6;73(11):e4568-e4577. doi: 10.1093/cid/ciaa752. PMID 32521007

RESULTS

PARTICIPANT FLOW:
Groups:
- Individualized Approach: The decolonization regimen will be performed only by those household members who experienced SSTI in the prior year.
  2% mupirocin ointment: Participants over 1 month of age, apply ointment to the anterior nares twice daily for 5 days.
  Bleach Bath (dilute): Participants over 1 month of age, pour 1/4 cup of bleach into a bath tub filled 1/4 full of water. Soak in bath for 15 minutes daily for 5 days.
  Hygiene Protocol: Follow key hygiene tips:
  * Throw out all lotions or creams that you dip your hands into and replace with pumps or pour bottles.
  * Use liquid(pour or pump) soaps instead of bar soaps.
  * Wash hands frequently or use hand sanitizer(with more than %60 alcohol) such as Germ-X or Purell.
  * Do not share personal care items such as razors, brushes, or deodorant.
  * Wash all sheets and towels in hot water. Wash sheets every week.
  * Use towels and wash cloths only once before washing and do not share.
- Household Approach: All members of the household will perform the decolonization regimen.
  2% mupirocin ointment: Participants over 1 month of age, apply ointment to the anterior nares twice daily for 5 days.
  Bleach Bath (dilute): Participants over 1 month of age, pour 1/4 cup of bleach into a bath tub filled 1/4 full of water. Soak in bath for 15 minutes daily for 5 days.
  Hygiene Protocol: Follow key hygiene tips:
  * Throw out all lotions or creams that you dip your hands into and replace with pumps or pour bottles.
  * Use liquid(pour or pump) soaps instead of bar soaps.
  * Wash hands frequently or use hand sanitizer(with more than %60 alcohol) such as Germ-X or Purell.
  * Do not share personal care items such as razors, brushes, or deodorant.
  * Wash all sheets and towels in hot water. Wash sheets every week.
  * Use towels and wash cloths only once before washing and do not share.
Period: Overall Study
Arm/Group | Individualized Approach | Household Approach
Started | 248 | 226
Completed | 218 | 199
Not Completed | 30 | 27
Not completed — Lost to Follow-up | 30 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individualized Approach | Household Approach | Total
Number analyzed (Participants) | 248 | 226 | 474
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 145 | 128 | 273
  Between 18 and 65 years | 101 | 97 | 198
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.65 (16.65) | 18.69 (15.94) | 18.67 (16.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 124 | 258
  Male | 114 | 102 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 13 | 29
  Not Hispanic or Latino | 232 | 213 | 445
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 59 | 126
  White | 169 | 162 | 331
  More than one race | 12 | 5 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 248 | 226 | 474
Height (inches) [Mean (Standard Deviation); unit: inches] | 54.95 (14.53) | 55.24 (15.80) | 55.09 (14.65)
Weight (pounds) [Mean (Standard Deviation); unit: pounds] | 114.09 (77.19) | 121.74 (88.25) | 117.85 (82.81)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of SSTI at 3 Months After Decolonization
Description: Cumulative Number of Participants with SSTI at any time during the 3 Months following Decolonization protocol
Time Frame: 3 months after enrollment
Population: 447 of 474 participants were analyzed. The remaining 27 participants were lost to follow up for this time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 235 | 212
Participants | 23 | 23
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.757, Fisher Exact

2. Secondary Outcome: Number of Participants With Incidence of SSTI at 1 Month After Decolonization
Description: Cumulative Number of Participants with SSTI at any time during the 1 Month following Decolonization protocol
Time Frame: 1 month after enrollment
Population: 449 of 474 participants were analyzed. The remaining 25 participants were lost to follow up for this time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 237 | 212
Participants | 8 | 8
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 1.00, Fisher Exact

3. Secondary Outcome: Number of Participants With Incidence of SSTI at 6 Months After Decolonization
Description: Cumulative Number of Participants with SSTI at any time during the 6 Months following Decolonization protocol
Time Frame: 6 months after enrollment
Population: 434 of 474 participants were analyzed. The remaining 40 participants were lost to follow up for this time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 225 | 209
Participants | 32 | 33
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.687, Fisher Exact

4. Secondary Outcome: Number of Participants With Incidence of SSTI at 9 Months After Decolonization
Description: Cumulative Number of Participants with SSTI at any time during the 9 Months following Decolonization protocol
Time Frame: 9 months after enrollment
Population: 433 of 474 participants were analyzed. The remaining 41 participants were lost to follow up for this time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 226 | 207
Participants | 39 | 35
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 1.00, Fisher Exact

5. Secondary Outcome: Number of Participants With Incidence of SSTI at 12 Months After Decolonization
Description: Cumulative Number of Participants with SSTI at any time during the 12 Months following Decolonization protocol
Time Frame: 12 months after enrollment
Population: 417 of 474 participants were analyzed. The remaining 57 participants were lost to follow up for this time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 218 | 199
Participants | 48 | 41
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.811, Fisher Exact

6. Secondary Outcome: Number of Participants Colonized With MRSA at 1 Month After Decolonization
Description: Number of Participants Colonized with MRSA at the 1 Month longitudinal study visit
Time Frame: 1 month after enrollment
Population: 438 of 474 participants were analyzed. The remaining 36 participants were lost to follow up for this time frame or were not available for swabs at the time of the home visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 230 | 208
Participants | 45 | 20
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.004, Fisher Exact

7. Secondary Outcome: Number of Participants Colonized With MRSA at 3 Months After Decolonization
Description: Number of Participants Colonized with MRSA at the 3 Month longitudinal study visit
Time Frame: 3 months after enrollment
Population: 433 of 474 participants were analyzed. The remaining 41 participants were lost to follow up for this time frame or were not available for swabs at the time of the home visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 224 | 209
Participants | 51 | 26
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.006, Fisher Exact

8. Secondary Outcome: Number of Participants Colonized With MRSA at 6 Months After Decolonization
Description: Number of Participants Colonized with MRSA at the 6 Month longitudinal study visit
Time Frame: 6 months after enrollment
Population: 431 of 474 participants were analyzed. The remaining 43 participants were lost to follow up for this time frame or were not available for swabs at the time of the home visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 227 | 204
Participants | 39 | 21
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.050, Fisher Exact

9. Secondary Outcome: Number of Participants Colonized With MRSA at 9 Months After Decolonization
Description: Number of Participants Colonized with MRSA at the 9 Month longitudinal study visit
Time Frame: 9 months after enrollment
Population: 422 of 474 participants were analyzed. The remaining 52 participants were lost to follow up for this time frame or were not available for swabs at the time of the home visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 226 | 196
Participants | 40 | 17
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.007, Fisher Exact

10. Secondary Outcome: Number of Participants Colonized With MRSA at 12 Months After Decolonization
Description: Number of Participants Colonized with MRSA at the 12 Month longitudinal study visit
Time Frame: 12 months after enrollment
Population: 407 of 474 participants were analyzed. The remaining 67 participants were lost to follow up for this time frame or were not available for swabs at the time of the home visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 215 | 192
Participants | 47 | 22
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.005, Fisher Exact

11. Secondary Outcome: Number of Participants Who Report Development of Adverse Effects Occurring During Decolonization Period
Description: Number of participants who report development of Nasal burning, itching, stinging, or runny nose or Skin itching, dry skin, or rash during the decolonization period.
Time Frame: 1 week after enrollment
Population: 309 participants were assigned decolonization measures as part of the protocol. Of these 11 participants were lost to follow-up and never returned their adherence documents. 4 participants did not complete any part of the assigned decolonization measures. The remaining 294 participants are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 84 | 210
Participants | 41 | 102
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Equivalence — testing equivalence of individualized approach compared to household approach; p = 1.00, Fisher Exact

12. Secondary Outcome: Number of All Recovered S. Aureus Isolates With High-level Mupirocin Resistance
Description: Number of all recovered S. aureus isolates resistant to mupirocin at the study visit before decolonization protocol and the study visit immediately after decolonization protocol
Time Frame: 1 month
Population: All participants swabbed before decolonization. 438 participants swabbed at 1 mo. follow-up (after decolonization) - remaining 36 lost to follow-up or unavailable for swabs at home visit. This SECONDARY outcome is independent of study group, as the impact of the study on mupirocin resistance in overall study population is the outcome measure.
Measure: Count of Units; unit: Isolates Analyzed/Recovered
Units Other Than Participants: Isolates Analyzed/Recovered
Groups:
- Before Decolonization: All isolates recovered across study before decolonization protocol began (enrollment visit)
- After Decolonization: All isolates recovered across study directly after decolonization protocol (1 month visit)
Arm/Group | Before Decolonization | After Decolonization
Number analyzed (Participants) | 474 | 438
Number analyzed (Isolates Analyzed/Recovered) | 808 | 492
Isolates Analyzed/Recovered | 31 | 20
Statistical Analysis 1: Comparison: Before Decolonization vs After Decolonization; Test type: Equivalence — testing equivalence of before and after decolonization protocol; p = 0.84, Chi-squared

13. Secondary Outcome: Number of Participants Incurring Economic Burden of Performing Protocol
Description: Number of participants incurring additional costs during their compliance with prescribed hygiene measures prescribed with the decolonization regimen: e.g., cost of containers of lotion or bars of soap discarded, cost of new pump or pour lotion or soap purchased, cost of new personal hygiene items or linens, cost of additional loads of laundry
Time Frame: 1 month after enrollment
Population: 435 of 474 participants returned their cost of protocol documentation. This SECONDARY outcome is independent of study group, as the economic impact of the study in the overall study population is the outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Entire Study Population: Additional costs of associated with protocol across all participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 435
Participants | 75

14. Secondary Outcome: Number of Participants Reporting a Confirmed MRSA Infection Over the 12-month Longitudinal Study Period.
Description: Number of participants reporting the development of a MRSA infection over the year of longitudinal follow-up that has been culture- and physician-confirmed through verification by medical record and culture report.
Time Frame: 1 Year
Population: 416 of 474 participants were analyzed. The remaining 58 participants were lost to follow up for this time frame and outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 218 | 198
Participants | 14 | 8
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Non-Inferiority — testing non-inferiority of individualized approach compared to household approach; p = 0.381, Fisher Exact

15. Secondary Outcome: Number of Participants Adhering to Decolonization Measures
Description: Number of participants Adhering to decolonization measures. Defined as reported completion of at least 4 of the 5 assigned days (8 or more mupirocin applications and 4 or more bleach baths)
Time Frame: 1 week
Population: 309 participants were assigned decolonization measures as part of the protocol. Of these 11 participants were lost to follow-up and never returned their adherence documents. The remaining 298 participants are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Approach | Household Approach
Number analyzed (Participants) | 86 | 212
Participants | 61 | 130
Statistical Analysis 1: Comparison: Individualized Approach vs Household Approach; Test type: Equivalence — testing equivalence of individualized approach compared to household approach; p = 0.143, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Individualized Approach | Household Approach
All-Cause Mortality (participants affected / at risk) | 0/248 | 0/226
Serious Adverse Events (participants affected / at risk) | 0/248 | 0/226
Other Adverse Events (participants affected / at risk) | 41/248 | 102/226
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Individualized Approach (N=248) | Household Approach (N=226)
Itching (from mupirocin) (General disorders) | 6 | 19
Runny nose (from mupirocin) (General disorders) | 11 | 30
Itching (from bleach baths) (General disorders) | 11 | 31
Dry skin (from bleach baths) (General disorders) | 24 | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT01814371/Prot_SAP_000.pdf